CLINICAL TRIAL: NCT01108562
Title: Treatment of Postoperative Pain After Total Hip Arthroplasty Using Intravenous Lidocaine Infusion in Combination With Patient Controlled Analgesia: a Prospective Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Treatment of Postoperative Pain After Total Hip Arthroplasty Using Intravenous Lidocaine Infusion
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Charles Lee MD (Unknown); Michelle Schlunt MD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 57366
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Postoperative Pain Management After Total Hip Arthroplasty
Keywords: postoperative pain management
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Patients will receive a Dilaudid PCA in combination with a placebo infusion of normal saline.
  Interventions: Other: Normal Saline
- Lidocaine Group (Experimental): Patients will be receive a Dilaudid PCA in combination with a continuous Lidocaine infusion.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Patients in the experimental group will be receiving a Lidocaine infusion at 1.33 mg/kg/hr for 24 hours postoperatively.
  Arms: Lidocaine Group
Other: Normal Saline — Patients in the control group will be receiving an infusion of normal saline for 24 hours postoperatively.
  Arms: Control Group

SUMMARY:
This study will focus on patients undergoing total hip arthroplasty and Loma Linda University Medical Center & East Campus. These patients will be randomized to receive a low dose lidocaine infusion or placebo, in addition to the patient controlled analgesia pump. These groups will be compared to one another statistically to determine which group shows the safest and most satisfying pain control.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female undergoing a total hip arthroplasty Subject is American Society of Anesthesiologists physical status 1, 2, or 3 Subject has voluntarily signed and dated the informed consent document approved by the IRB Be English speaking

Exclusion Criteria:

* Age > 80 years old or younger than 18 years old Congestive heart failure Hepatic insufficiency Neurological disorders Psychiatric disorders Steroid treatment No history of atrial fibrillation Chronic pain disorder with opioid treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
We propose to test the hypothesis that adding a low dose lidocaine infusion to patient controlled analgesia will lower the amount of opioids that these patients will receive, thereby improving patient safety while still providing adequate analgesia. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Schlunt, MD, Principal Investigator — Loma Linda University Medical Center